CLINICAL TRIAL: NCT01191424
Title: A Multicenter, Multinational, Single-Dose, Open Label, Randomized, 2-Way Crossover, Clinical Pharmacology Study of CHF 1535 100/6 Next™ DPI (Fixed Combination of Beclomethasone Dipropionate 100 µg Plus Formoterol 6 µg) Versus the Free Combination of Licensed Beclomethasone DPI and Formoterol DPI in Asthmatic Adolescents and Adult Patients
Brief Title: A Study Comparing the Pharmacokinetic, Pharmacodynamic and Safety of CHF 1535 (Fixed Combination of Beclomethasone + Formoterol) Administered Via the NEXT DPI, Versus the Free Combination of Licenced Beclomethasone DPI and Formoterol DPI in Asthmatic Adolescent and Adult Patients.
Acronym: ADONE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCD-1017-PR-0034; 2010-018947-33 (EudraCT Number)
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Asthma
Keywords: Asthma; PK; Adolescents; Adults
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHF1535 NEXT DPI (Experimental): Male and female adolescents and adult patients (≥ 12 years old) treated with CHF1535 NEXT DPI
  Interventions: Drug: CHF1535 NEXT DPI
- Free combination BDP and FF (Active Comparator): Male and female adolescents and adult patients (≥ 12 years old) treated with a free combination of licenced BDP and FF
  Interventions: Drug: BDP DPI and formoterol DPI

INTERVENTIONS:
Drug: CHF1535 NEXT DPI — FIXED COMBINATION OF BECLOMETHASONE DIPROPIONATE 100µg PLUS FORMOTEROL FUMARATE 6 µg DRY POWDER INHALER
  Arms: CHF1535 NEXT DPI
Drug: BDP DPI and formoterol DPI — FREE COMBINATION OF LICENSED BECLOMETHASONE DPI AND FORMOTEROL DPI
  Arms: Free combination BDP and FF

SUMMARY:
The purpose of this study is to demonstrate that the CHF 1535 (fixed combination of Beclometasone Dipropionate (BDP) 100 µg / Formoterol Fumarate (FF) 6 µg) delivered via the NEXT Dry Powder Inhaler (DPI) does not show a greater exposure to BDP, Beclometasone-17-Monopropionate(B17MP, active metabolite of BDP) and FF in comparison to a free combination of BDP DPI plus FF DPI licensed products after a morning dose administration of BDP and FF (total dose of BDP 400 µg / FF 24 µg) in adolescent and adult asthmatic patients.

ELIGIBILITY:
Main Inclusion Criteria:

1. Male and female adolescents (≥ 12 years old) and adults (≥18 and ≤ 65 years old)
2. Written informed consent;
3. Diagnosis of asthma as defined in the GINA guidelines;
4. Patients with stable asthma, according to the Investigator's opinion;
5. Asthmatic patients already treated with ICS or using short-acting inhaled β2-agonists as reliever to control asthma symptoms;
6. Patients with a forced expiratory volume in one second (FEV1) > 70% of predicted values;
7. Patients with a peak inspiratory flow (PIF) > 40 L/min
8. Reversibility test;
9. Non- or ex-smokers;
10. A cooperative attitude and ability to be trained about the proper use of DPI and compliant to study procedures;

Main Exclusion Criteria:

1. Pregnant or lactating female;
2. Having received an investigational drug within 2 months before the screening visit
3. Diagnosis of COPD as defined by the current GOLD guidelines;
4. Significant medical history of and/or treatments for cardiac, renal, neurological, hepatic, endocrine diseases, or any laboratory abnormality;
5. Known hypersensitivity to the active treatments;
6. History of drug addiction or excessive use of alcohol;
7. Treatment with a xanthine derivative (e.g. theophylline) formulation in the 4 weeks prior to screening;
8. Hospitalization due to asthma exacerbation or asthma exacerbation within 1 month prior to the screening visit;
9. Inability to perform the required breathing technique and blood sampling;
10. Lower respiratory tract infection within 1 month prior to the screening visit;
11. Blood donation (450 mL or more) or significant blood loss in the 12 weeks before the screening visit.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Systemic exposure to B17MP (active metabolite of BDP) after single dose (4 inhalations) of CHF1535 100/6 NEXT DPI in comparison with an already approved free combination of BDP DPI and FF DPI | 0-8hrs
  Plasma AUC0-t for B17MP

SECONDARY OUTCOMES:
Different pharmacokinetic parameters | 0-8hrs
  BDP/B17MP and FF PK parameters
Lung function parameters | 0-8hrs
  Peak FEV1, FEV1 time averaged value (FEV1 AUC0-t/8).
Plasma potassium | 0-8hrs
  Plasma Potassium Cmin, tmin and AUC0-t
Plasma glucose | 0-8hrs
  Plasma Glucose Cmax, tmax, AUC0-2h and AUC0-t
Heart rate | 0-8hrs
  time averaged value (AUC0-t/8)
Adverse Events | during the whole study period

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Study Director — Medicines Evaluation Unit; Hans Bisgaard, MD, Study Director — Copenhagen University Hospital at Herlev
Locations (2):
- Copenhagen University Hospital, Copenhagen, Denmark
- Medicines Evaluation Unit, Manchester, United Kingdom

REFERENCES:
- [Background] Govoni M, Piccinno A, Lucci G, Poli G, Acerbi D, Baronio R, Singh D, Kuna P, Chawes BL, Bisgaard H. The systemic exposure to inhaled beclometasone/formoterol pMDI with valved holding chamber is independent of age and body size. Pulm Pharmacol Ther. 2015 Feb;30:102-9. doi: 10.1016/j.pupt.2014.04.003. Epub 2014 Apr 16. PMID 24746942
- [Result] Chawes BL, Govoni M, Piccinno A, Kreiner-Moller E, Vissing NH, Mortensen L, Nilsson E, Bisgaard A, Deleuran M, Skytt N, Samandari N, Acerbi D, Bisgaard H. A clinical pharmacology study of fixed vs. free combination of inhaled beclometasone dipropionate and formoterol fumarate dry powder inhalers in asthmatic adolescents. Br J Clin Pharmacol. 2014 Nov;78(5):1169-71. doi: 10.1111/bcp.12424. No abstract available. PMID 24830339
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2010-018947-33